CLINICAL TRIAL: NCT07007065
Title: A Randomized, Controlled, Partially Masked, Phase 3b Study to Assess the Injection Burden, Efficacy, Safety, and Long-Term Preservation of Visual Acuity of Surabgene Lomparvovec (ABBV-RGX-314) in a Real-World Context in Subjects With Neovascular Age-Related Macular Degeneration (nAMD)
Brief Title: Study to Assess the Injection Burden, Adverse Events, Change in Disease Activity, and Long-Term Preservation of Visual Acuity of Surabgene Lomparvovec in Adult Participants With Neovascular Age-Related Macular Degeneration (nAMD)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M24-528; 2024-512298-28-00 (Other: EU CT)
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: Neovascular age-related macular degeneration; Surabgene Lomparvovec; ABBV-RGX-314

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Surabgene Lomparvovec (ABBV-RGX-314) Dose 1 (Experimental): Participants will receive Surabgene Lomparvovec (ABBV-RGX-314) Dose 1 administered via subretinal delivery one time.
  Interventions: Drug: Surabgene Lomparvovec (ABBV-RGX-314)
- Surabgene Lomparvovec (ABBV-RGX-314) Dose 2 (Experimental): Participants will receive Surabgene Lomparvovec (ABBV-RGX-314) Dose 2 administered via subretinal delivery one time.
  Interventions: Drug: Surabgene Lomparvovec (ABBV-RGX-314)
- Ranibizumab Control Group (Experimental): Ranibizumab administered via intravitreal injection as needed PRN
  Interventions: Drug: Ranibizumab Control

INTERVENTIONS:
Drug: Surabgene Lomparvovec (ABBV-RGX-314) — subretinal injection
  Other Names: Surabgene Lomparvovec
  Arms: Surabgene Lomparvovec (ABBV-RGX-314) Dose 1; Surabgene Lomparvovec (ABBV-RGX-314) Dose 2
Drug: Ranibizumab Control — intravitreal injection
  Arms: Ranibizumab Control Group

SUMMARY:
Neovascular age-related macular degeneration (nAMD), also known as "wet" AMD, is the abnormal growth of new blood vessels in the light-sensitive tissue at the back of the eye called the retina. The purpose of this study is to assess how safe and effective Surabgene Lomparvovec is in treating participants with Neovascular age-related macular degeneration (nAMD).

Surabgene Lomparvovec (ABBV-RGX-314) is an investigational gene therapy being developed for the treatment of neovascular age-related macular degeneration (nAMD). Participants will be placed into 1 of 3 groups, called treatment arms. Each group receives different treatment. Adult participants aged 50 and older years with a diagnosis of previously treated nAMD will be enrolled. Around 561 participants will be enrolled in the study at approximately 150 sites worldwide.

Participants in groups 1 and 2 will receive a single subretinal dose of ABBV-RGX-314. Participants in group 3 will receive Ranibizumab as needed throughout the study. Ranibizumab will be given as an intravitreal injection (injection into the jelly-like tissue that fills the eyeball injection), and ABBV-RGX-314 will be given as a subretinal (between the retina and the back of the eye) injection. The Assessment Period begins after randomization (1:1:1) to one of the ABBV-RGX-314 treatment groups or control at Week -2 and lasts up to 5 years.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular monthly visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Pseudophakic (at least 12 weeks post cataract surgery at Screening Visit 1 [Week -6]) in the study eye.
* Must have a diagnosis of choroidal neovascularization (CNV) secondary to age-related macular degeneration (AMD) in the study eye

  --CNV lesion characteristics as assessed by the central reading center: lesion size needs to be less than 10-disc areas (typical disc area = 2.54 mm^2)
* Must have received at least 2 intravitreal anti-vascular endothelial growth factor (VEGF) injections in the past 6 months in the study eye prior to Screening Visit 1 (Week -6) and have been responsive (determined by investigator)

Exclusion Criteria:

* CNV or macular edema in the study eye that is secondary to any causes other than AMD
* Study eye with nAMD diagnosed > 4 years from Screening Visit 1
* Any retinal pigment epithelial detachment > 400 μm or any pigment epithelial detachment > 350 μm within the central subfield (central 1 mm) in the study eye at Screening Visit 1 (Week -6), as assessed by the central reading center.
* Any subretinal hemorrhage in the study eye > 50% of the total lesion area or within the parafovea (3 mm center of the macula), as determined by the central reading center
* Retinal pigment epithelial tear involving the central subfield (central 1 mm) in the study eye as determined by the central reading center.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 561 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2033-03 (Estimated); Study Completion 2033-03 (Estimated)

PRIMARY OUTCOMES:
Annualized intravitreal anti-VEGF injection rate | Up to Week 54
  To assess the injection burden and the necessity for supplemental anti-VEGF injections over the first year of the study period across the different treatment groups.
Number of Participants Experiencing Adverse Events | Up to 5 years
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Change from Baseline in best corrected visual acuity (BCVA) | Up to 3 Years
  BCVA will be measured using an Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart
Annualized intravitreal anti-VEGF injection rate | Up to 3 Years
  To evaluate the long-term injection burden and the necessity for supplemental anti-VEGF injections across the different treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (44):
- United States (24):
  - American Vision Partners /ID# 264615, Sun City, Arizona
  - Retinal Diagnostic Center /ID# 263054, Campbell, California
  - The Retina Partners /ID# 263265, Encino, California
  - Retinal Consultants - Sacramento - Greenback Lane /ID# 263983, Sacramento, California
  - Retina Consultants of Southern Colorado /ID# 263284, Colorado Springs, Colorado
  - Colorado Retina Associates /ID# 263247, Lakewood, Colorado
  - Advanced Vision Surgery Center /ID# 264208, Longmont, Colorado
  - Advanced Research, LLC /ID# 276526, Deerfield Beach, Florida
  - Retina Vitreous Consultants LLP business DBA as Retina Group of Florida /ID# 264631, Fort Myers, Florida
  - Florida Retina Institute - Lake Mary /ID# 263288, Lake Mary, Florida
  - Southeast Retina Center /ID# 263264, Augusta, Georgia
  - Springfield Clinic Main Campus /ID# 265202, Springfield, Illinois
  - Wolfe Eye Clinic - West Des Moines /ID# 263270, West Des Moines, Iowa
  - The Retina Care Center /ID# 263263, Baltimore, Maryland
  - Retina Specialist /ID# 264633, Towson, Maryland
  - Associated Retinal Consultants /ID# 263289, Royal Oak, Michigan
  - Erie Retina Research /ID# 263287, Erie, Pennsylvania
  - Charleston Neuroscience Institute /ID# 264037, Bluffton, South Carolina
  - Charleston Neuroscience Institute /ID# 276425, Charleston, South Carolina
  - Retina Consultants of South Carolina - Ladson /ID# 277596, Ladson, South Carolina
  - Retina Consultants of America /ID# 264038, Mt. Pleasant, South Carolina
  - Austin Clinical Research, LLC /ID# 263229, Austin, Texas
  - Star Retina - Burleson /ID# 266386, Burleson, Texas
  - Retina Consultants of Texas - Westover /ID# 264209, San Antonio, Texas
- Austria (2):
  - Medizinische Universitaet Innsbruck /ID# 264502, Innsbruck, Tyrol
  - Kepler Universitaetsklinikum GmbH /ID# 264493, Linz, Upper Austria
- Medical Center -Vereya /ID# 275728, Stara Zagora, Bulgaria
- Retina Centre of Ottawa /ID# 263803, Ottawa, Ontario, Canada
- France (3):
  - Hopital Edouard Herriot /ID# 265072, Lyon, Auvergne-Rhône-Alpes
  - Centre Hospitalier Universitaire de Nantes - L' Hopital l'hôtel-Dieu /ID# 265077, Nantes, Pays de la Loire Region
  - Centre Hospitalier Intercommunal de Creteil /ID# 265080, Créteil, Val-de-Marne
- Germany (5):
  - Universitaetsklinikum Freiburg /ID# 275449, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen /ID# 264283, Tübingen, Baden-Wurttemberg
  - Universitaetsklinikum Bonn /ID# 264279, Bonn, North Rhine-Westphalia
  - Universitaetsklinikum Schleswig-Holstein - Campus Luebeck /ID# 264284, Lübeck, Schleswig-Holstein
  - Universitaetsklinikum Hamburg-Eppendorf /ID# 264280, Hamburg
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Universita Cattolica /ID# 276032, Rome, Roma, Italy
- Spain (3):
  - Hospital Universitario Puerta de Hierro - Majadahonda /ID# 263179, Majadahonda, Madrid
  - Institut Clínic d'Oftalmologia (ICOF). Hospital Clínic d'Oftalmologia. /ID# 263152, Barcelona
  - Hospital Universitario 12 de Octubre /ID# 263544, Madrid
- United Kingdom (4):
  - Gloucestershire Royal Hospital /ID# 276072, Gloucester, Gloucestershire
  - The Retina Clinic London /ID# 266156, London, Greater London
  - Liverpool University Hospitals NHS Foundation Trust /ID# 265854, Liverpool, Merseyside
  - Bristol Eye Hospital /ID# 266155, Bristol

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-528